CLINICAL TRIAL: NCT06531473
Title: Laser Outcomes Associated With HoLEP Procedures
Brief Title: Laser Outcomes Associated With (Holmium Laser Enucleation of the Prostate) HoLEP Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Urologic Surgeon, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00220458
Record Dates: First submitted 2024-06-26; First posted 2024-08-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Urologic Diseases; Prostate Obstruction
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2J 40hz Laser Energy (Experimental): Patients will under go their Holmium Laser Enucleation procedure with the laser setting: 2J 40hz
  Interventions: Procedure: HoLEP
- 2J 50hz Laser Energy (Experimental): Patients will under go their Holmium Laser Enucleation procedure with the laser setting: 2J 50hz
  Interventions: Procedure: HoLEP
- 2J 60hz Laser Energy (Experimental): Patients will under go their Holmium Laser Enucleation procedure with the laser setting: 2J 60hz
  Interventions: Procedure: HoLEP

INTERVENTIONS:
Procedure: HoLEP — Patients will be randomized to one of the laser energy groups day of surgery.

SUMMARY:
The primary aim is to assess the impact of laser setting frequency and wattage during holmium laser enucleation of the prostate. There is currently no gold-standard laser settings for HoLEP procedures. In the investigator's current high-volume practice, the following settings for enucleation are: 2j 50hz. These settings are conventional settings, but there is no literature to prove optimal laser settings. The investigators hypothesizes that utilization of higher laser settings may be associated with a clinically significant (defined as > 10%) decrease in procedural time without any detrimental postoperative outcomes, and a utilization of lower laser settings may be associated with a clinically significant (defined as >10%) reduction in postoperative irritative voiding symptoms without any detrimental postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males 18-89 who are undergoing HoLEP for the treatment of bothersome lower urinary tract symptoms, that are typically caused by enlarged prostates

Exclusion Criteria:

* Prostates measurements over 200g
* Patients who lack decisional capacity
* Patients who are non-english speakers

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Identifying Outcomes of 40 hz, 50 hz and 60 hz laser setting groups during Holmium Laser Enucleation of the Prostate. | 2 years
  Comparing operative outcomes between the 40 hz, 50 hz and 60 hz laser setting groups.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Krambeck, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No